CLINICAL TRIAL: NCT02822456
Title: Intermittent Oro-Esophageal Tube Feeding Using Individually-Customized 3-Dimensional Printing: Prospective, Single Center, Observational Trial of Superiority
Brief Title: Intermittent Oro-Esophageal Tube Feeding Using Individually-Customized 3-Dimensional Printing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate Professor, Ulsan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chhwang5
Record Dates: First submitted 2016-06-14; First posted 2016-07-04 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Dysphagia
Keywords: dysphagia; intermittent tube; individual 3D printed guiding tube
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individual 3D-printed guided tube (Experimental): IOE tube feeding using individual 3D-printed guided tube and nelaton tube whenever they eat
  Interventions: Procedure: VFSS
- traditional IOE tube (Active Comparator): classic IOE tube feeding using nelaton tube only whenever they eat
  Interventions: Procedure: VFSS
- nasogastric tube (Active Comparator): nasogastric tube feeding using levin tube always
  Interventions: Procedure: VFSS

INTERVENTIONS:
Procedure: VFSS — VFSS using assignment of tube type among the interventions such as individual 3D printed guiding tube, traditional IOE tube, levin tube

SUMMARY:
The aim of this study is to test the clinical effectiveness of IOE tube using individually customized 3-dimentional printed guiding tube as an alternative to Levin tube feeding when unconscious patients have no choice but tube feeding.

DETAILED DESCRIPTION:
According to standard Guideine of videofluoroscopic swallow study(VFSS), Patients referred to dysphagia(swallowing dysfunction)who were required to tube feeding and medically stable of vital sign, and agreed to participate. Participants with swallowing dysfunction who were classified into three groups (nasogastric tube, traditional intermittent (IOE) tube, individual 3D printed guiding tube) according to VFSS.

Both traditional IOE tube and individual 3D printed guiding tube groups will receive training about procedure prior to the first feeding. All participants will be evaluated with satisfaction for tube feeding (EORTC QLQ-H&N35) in 3 days from the start day of the tube feeding. On the day of oral feeding, participants will be evaluated with the questionnaires and clinical examination. If the participant is discharged in a state maintain the tube feeding, investigated further length stay at leaving the hospital. On the 1 month, 3 month from tube feeding, the investigators will follow-up and measure the questionnaires and clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Dysphagia patients to check in VFSS (videofluoroscopic swallow study)
* Patients participating in the study agreement
* Oral feeding is not possible (Need tube feeding)

Exclusion Criteria:

* Patient to reject the participation
* Crico-pharyngeal incoordination
* Impaired esophageal peristalsis
* Impaired GI tract
* Observed esophageal reflux

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change of EORTC QLQ - H&N35 index | 1 month after start of tube feeding
  Details (inconvenience, discomfort, altered body image, social activities, family life, pain, ease of learning to use) satisfaction evaluation (3, 9, 10)

SECONDARY OUTCOMES:
complications | after 1st session (3days) and after 1 month, and after 3 months
  whether aspiration pneumonia on Chest Radiography or not, Measurement at leave hospital or start oral feeding can be another endpoint
change Mid-arm circumference | before VFSS and 1 month and 3 months after start of tube feeding
change of Serum albumin | before VFSS and 1 month and 3 months after start of tube feeding
change of MRS index | before VFSS and 1 month and 3 months after start of tube feeding
change of success rate (rate of elimination) | after 1st session (3days), after 1 month, and after 3 months
change of EORTC QLQ - H&N35 index | after 1st session (3days) and after 3 months
  Measurement at leave hospital or start oral feeding can be another endpoint, Details (inconvenience, discomfort, altered body image, social activities, family life, pain, ease of learning to use) satisfaction evaluation (3, 9, 10)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No